CLINICAL TRIAL: NCT03232242
Title: Application of Next Generation Sequencing Technique in Precise Diagnosis of Infectious Diseases
Brief Title: Application of NGS Technique in Precise Diagnosis of Infectious Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director, Huashan Hospital
Other Study IDs: KY2017-338
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Next Generation Sequencing; Infectious Disease
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Next-generation sequencing — To provide rapid etiological diagnosis of patients by means of next-generation sequencing.

SUMMARY:
Infectious disease leads to deaths that accounted for more than 25% of all causes of human mortality. But the traditional microbiological diagnostic methods such as specimen culture are sometimes time-consuming, and have limited sensitivity. And some bacteria, anaerobes and viruses may be difficult to cultivate and isolation. Therefore, the accurate identification and rapid classification of pathogenic microorganisms is very important for the patient's precise diagnosis and timely treatment.

Small-scale studies on the diagnostic efficacy and prognosis of infection in the next generation have been shown to provide early diagnosis and targeted medication guidance for bloodstream infections and respiratory infections, but the larger-scale validation of next-generation sequencing Technology in the diagnosis and treatment of infectious diseases in the human body is relatively rare.

The purpose of this study is to provide rapid etiological diagnosis of patients by means of next-generation sequencing, to change the way of treatment of patients under the existing traditional pathogen detection by means of accurate description of pathogens and monitoring their dynamic changes, and to provide patients with more accurate treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients are highly suspected of fever of unknown origin
* Patients are highly suspected of bloodstream infection
* Patients are highly suspected of respiratory infections
* Patients are highly suspected of central nervous system infection

Exclusion Criteria:

* Patients diagnosed as non-infectious diseases such as cancer and autoimmune diseases;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are highly suspected of infectious diseases, and they will be selected mainly from infectious diseases departments .
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value (sensitivity and sensibility, positive/negative predictive value) of next-generation sequencing in the pathogen detection of infectious diseases | 3 years
  We aim to collect samples from patients with fever, bacteremia and bloodstream infections, respiratory infections, central nervous system infections, and abscesses, including blood, cerebrospinal fluid, serous effusion, pus, sputum, alveolar lavage fluid, throat swab. Next-generation sequencing will be performed on the collected samples. Our analysis of the sequencing results will focus on the analysis and identification of pathogen genes and will compare the diagnostic performance of next-generation sequencing with conventional etiological diagnostic methods. We anticipate that next-generation sequencing in infectious patients will show a greater diagnostic value than the traditional methods (including culture, special pathogen serology, PCR detection of nucleic acids, etc.).

SECONDARY OUTCOMES:
Diagnostic value (sensitivity and sensibility, positive/negative predictive value) of traditional methods in the pathogen detection of infectious diseases | 3 years
  We aim to collect samples from patients with fever, bacteremia and bloodstream infections, respiratory infections, central nervous system infections, and abscesses, including blood, cerebrospinal fluid, serous effusion, pus, sputum, alveolar lavage fluid, throat swab. Traditional methods including culture, special pathogen serology, PCR detection of nucleic acids, etc, will be performed on the collected samples. Our analysis aims to study the diagnostic power of the traditional diagnostic methods in infectious diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fu Z, Ai J, Zhang H, Cui P, Xu T, Zhang Y, Zhang Y, Wu H, Shen A, Lin K, Zhang M, Qiu C, Jiang N, Zhou Y, Zhang W. Pathogen quantitative efficacy of different spike-in internal controls and clinical application in central nervous system infection with metagenomic sequencing. Microbiol Spectr. 2023 Dec 12;11(6):e0113923. doi: 10.1128/spectrum.01139-23. Epub 2023 Nov 20. PMID 37982612